CLINICAL TRIAL: NCT01217996
Title: Computerized Intervention for Amelioration of Cognitive Late Effects Among Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COGTRN; 120421-RSGPB-11-009-01-CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Brain Tumor; Acute Lymphoblastic Leukemia
Keywords: working memory intervention; memory impairment; cognitive late effects; Childhood Cancer Survivors
MeSH Terms: conditions — Brain Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Memory Disorders | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Other): Children treated for a brain tumor (BT) or acute lymphoblastic leukemia (ALL) will complete the computerized working memory training program (intervention).
  Interventions: Behavioral: Computerized working memory training program (intervention)
- Control Group (Other): Children treated for a brain tumor (BT) or acute lymphoblastic leukemia (ALL) will complete the computerized working memory training program (control).
  Interventions: Behavioral: Computerized working memory training program (control)

INTERVENTIONS:
Behavioral: Computerized working memory training program (intervention) — A computer-based training program will be completed in the home. This program requires approximately 30 minutes every weekday for five weeks. The program software guides the child through eight rotating exercises each day, with increasing difficulty based on the child's level of performance. Exercises train both visuospatial and verbal WM using child-friendly activities. A research team member will serve as a coach who monitors weekly progress online and offers support through weekly phone calls with the study participants and their caregivers). Intervention participants will also partake in neuroimaging exams before and after the intervention
  Arms: Intervention Group
Behavioral: Computerized working memory training program (control) — Participants randomized to the control group will not complete any intervention during the intervention time period and will not partake in neuroimaging exams. They will complete an immediate and six month post follow-up cognitive assessment. Following completion of these assessments, they will be provided the opportunity to complete the computer-based training program off study.
  Arms: Control Group

SUMMARY:
Children treated for a brain tumor (BT) or acute lymphoblastic leukemia (ALL) show elevated rates of working memory impairment. Working memory (WM) is the ability to hold and manipulate information online; for example, when an individual mentally rehearses a phone number in order to dial it without writing it down. A computer-based working memory intervention has been successful in children diagnosed with ADHD and stroke survivors. Individuals participating in the intervention showed improvements on working memory measures as well as more complex problem solving skills. Neuroimaging (brain scans) conducted before and after training showed changes in brain activation suggestive of underlying changes in brain systems that support working memory. This study investigates the effectiveness of this computer-based working memory intervention for childhood cancer survivors.

DETAILED DESCRIPTION:
Participants randomized to the intervention arm will complete the computerized working memory training program. This computer-based training program is completed in the home and requires approximately 30 minutes every weekday for five weeks. The program software guides the child through eight rotating exercises each day, with increasing difficulty based on the child's level of performance. Exercises train both visuospatial and verbal WM using child-friendly activities. A research team member will serve as a coach who monitors weekly progress online and offers support through weekly phone calls with the study participants and their caregivers. This individual will not complete post-intervention assessments to maintain study blind. A home computer with internet connection and speakers is required. A laptop computer and/or wireless internet access will be provided to families whose only obstacle to participation is lack of computer access or internet connectivity in the home setting. Families randomized to the WM intervention will complete a tutorial with study staff that provides instruction in using a computer, the internet and the WM training software.

The objective of this study is to investigate the benefits of this working memory intervention in a sample of childhood cancer survivors and look at brain-based changes that may occur as the result of working memory intervention. To achieve this goal, we plan to study childhood cancer survivors randomly assigned to the working memory intervention or a passive waitlist. Both groups will participate in cognitive testing pre-, post-, and six months post intervention. Intervention participants will also partake in neuroimaging exams before and after the intervention. Findings from this study have direct potential to support a nonpharmaceutical cognitive intervention for cancer survivors that is a safe and effective alternative to stimulant medications with great promise for improving quality of life.

ELIGIBILITY:
Inclusion Criteria for Screening Phase:

* Received CNS-directed treatment (intrathecal chemotherapy or cranial irradiation) for a BT or ALL
* Infratentorial tumor location (for the BT cohort)
* Off treatment for at least one year with no evidence of recurrent or progressive disease
* Age 8-16 years inclusive at the time of enrollment
* English as the primary language
* Research participant and one parent willing to participate and provide consent/assent according to institutional guidelines

Exclusion Criteria for Screening Phase

* Significant impairment in global intellectual functioning (estimated or full scale IQ < 70 based on standardized testing routinely conducted on primary treatment protocols)
* History of CNS injury/disease predating or unrelated to cancer diagnosis
* Documented ADHD predating cancer diagnosis
* Treatment with psychostimulant or psychotropic medication within two weeks of study participation
* Major sensory or motor impairment that would preclude valid cognitive testing secondary to inability to complete study procedures (e.g., blindness, paresis, poorly controlled seizures/photosensitive epilepsy, psychosis)

Inclusion Criteria for Intervention Phase

* Signed screening consents and has undergone screening
* Fully evaluable psychological testing results (including IQ > or = 70)
* Age-scaled score on Digit Span, Letter-Number Sequencing or Spatial Span < 7 OR at least one standard deviation below IQ score
* Training aide is available to participate in required sessions
* Participant and training aide demonstrate computer proficiency
* Participant has access to or will be provided a laptop or home computer with internet connection and speakers
* Participant willing to participate in required aspects of computerized intervention
* Participant is able to take part in fMRI without sedation

Exclusion Criteria for Intervention Phase

* Major psychological condition that would preclude completion of protocol intervention (e.g., significant oppositionality, autism spectrum disorder, severe anxiety or depressive symptoms)
* Orthodontic appliances that cause MRI distortion or signal loss outside the mouth and sinus area

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
This study will measure working memory, attention and executive functions | Baseline, 10 weeks, and 6 months
  Participants in the working memory intervention will demonstrate significantly greater improvement from pre- to immediate post-intervention on performance- and rater-based measures of working memory relative to childhood cancer survivors placed on an intervention waitlist.

SECONDARY OUTCOMES:
The study will measure the maintenance of improvements on measures of working memory, attention and executive functions | 6 months.
  The improvements will be evaluated at six months following participation in the computer-based intervention program.
This study will examine the neural correlates of working memory before and immediately after intervention | Baseline and 10 weeks.
  This objective will use fMRI to examine the neural correlates of working memory before and immediately after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Conklin, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org